CLINICAL TRIAL: NCT03183011
Title: Cardiac Magnetic Resonance Imaging After Cardiac Resynchronization Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kenneth Bilchick, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Bilchick, MD, Associate Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRIPOSTCRT
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure, Systolic
Keywords: cardiac resynchronization therapy; implantable cardioverter defibrillator; heart failure; magnetic resonance imaging
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-CRT MRI (Other): This study has a single arm. Enrolled patients will follow the protocol as described, including evaluation with MRI, echocardiography, and cardiopulmonary exercise testing.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Cardiac MRI

SUMMARY:
This study is evaluating how MRI after CRT can provide key insights regarding LV function, structure, and mechanics resulting from CRT in patients with or without LV scar and inform optimal pacing strategies. The expected accurate and reproducible response assessment with cardiac MRI has important implications for evaluating CRT outcomes in clinical trials, and the insights from the post-CRT MRI promise to improve implementation of CRT.

DETAILED DESCRIPTION:
We are performing a study of 40 patients with current accepted indications for CRT and no MRI contraindications. These patients will have a pre-CRT MRI and another post-CRT MRI 6 months after the CRT procedure. Echocardiography, cardiopulmonary exercise testing, symptom assessment, and laboratory testing are also performed before and after CRT. Modifications to the post-CRT MRI protocol include the use of gradient echo cine imaging rather than steady state free precession imaging, application of wideband imaging to the LGE acquisitions, and strain imaging with cine Displacement Encoding with Stimulated Echoes (DENSE) tailored for device patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic systolic HF
* LVEF 35% or less
* Guideline-based class I or IIa indication for CRT
* 25 and 85 years old
* Predominantly in sinus rhythm
* GFR ≥ 40 ml/min/1.73m2* *Contrast will not be given for the 6-month follow-up scan if the GFR falls to < 40 ml/min/1.73m2.

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Presence of metal embedded in the body due to prior accident or injury, as documented by skull films or other imaging
* Preexisting pacemaker or defibrillator prior to enrollment
* Cerebral aneurysm clips; 6) cochlear implants
* Other metallic implants (prior to enrollment) known to be contraindications to MRI
* Severe claustrophobia
* Acute kidney injury
* Acute renal failure or chronic kidney disease with GFR < 40 cc/min
* Liver transplant
* Gadolinium allergy

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
CRT Response | 1 year
  CRT Response

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Bilchick, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auger DA, Bilchick KC, Gonzalez JA, Cui SX, Holmes JW, Kramer CM, Salerno M, Epstein FH. Imaging left-ventricular mechanical activation in heart failure patients using cine DENSE MRI: Validation and implications for cardiac resynchronization therapy. J Magn Reson Imaging. 2017 Sep;46(3):887-896. doi: 10.1002/jmri.25613. Epub 2017 Jan 9. PMID 28067978
- [Background] Ramachandran R, Chen X, Kramer CM, Epstein FH, Bilchick KC. Singular Value Decomposition Applied to Cardiac Strain from MR Imaging for Selection of Optimal Cardiac Resynchronization Therapy Candidates. Radiology. 2015 May;275(2):413-20. doi: 10.1148/radiol.14141578. Epub 2015 Jan 9. PMID 25581423